CLINICAL TRIAL: NCT05993169
Title: Body Composition Optimization Intervention to Increase Conversion to Surgical Candidacy: A Randomized Controlled Trial
Brief Title: Body Composition Optimization Intervention RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of feasibility.
Sponsor: Jacob M. Elkins (Other)
Responsible Party: Sponsor-Investigator, Jacob M. Elkins, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202306474
Record Dates: First submitted 2023-08-02; First posted 2023-08-15 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Primary care provider will be blind to subject arm,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Normal Care
- Nutritional consultation (Experimental): Patients who are selected into the body composition optimization (BCO) visits group will attend an extra one hour in-person check-up with Olivia Johnson as part of their regular clinic follow-ups. During their initial BCO visit, patients will complete a hard copy intake form. These BCO visits will take place in the same clinic as the regular visits. These visits will focus on individual concerns and goal-setting. These visits may be changed to online/video follow ups if the patients are finding it difficult to return to main campus that often.
  Interventions: Other: Body Composition optimization visits

INTERVENTIONS:
Other: Body Composition optimization visits — Patients who are selected into the body composition optimization (BCO) visits group will attend an extra one hour in-person check-up with Olivia Johnson as part of their regular clinic follow-ups. During their initial BCO visit, patients will complete a hard copy intake form. These BCO visits will take place in the same clinic as the regular visits. These visits will focus on individual concerns and goal-setting. These visits may be changed to online/video follow ups if the patients are finding it difficult to return to main campus that often.
  Arms: Nutritional consultation

SUMMARY:
This study aims to identify if the addition of structured nutrition/weight loss counseling to patients at the bariatric clinic can increase the conversion from bariatric clinic to surgical candidacy from (the current) 11% to a goal of 20% by way of tracking their BIA measurements.

DETAILED DESCRIPTION:
Obesity, at a BMI exceeding 40kg/m2 (class III) obesity, is a major risk factor for osteoarthritis (OA). In arthroplasty (joint replacement), patients in this population are routinely turned away due to surgeons refusing surgical treatment in patients above arbitrary BMI thresholds (typically 35 or 40 kg/m2). Due to this, patients often turn to simple weight loss to fall below these thresholds. Simple weight loss, which can include loss of muscle mass, has been proven ineffective, counterproductive, and to be an additional risk factor for surgery. To combat this, efforts in our dedicated bariatric clinic have been made to encourage muscle mass gain and body fat loss over simple weight loss methods where progress has been tracked through stationary, multi-frequency bioimpedance analysis (BIA). BIA is a readily available technology offered to industry and consumers. Our department is a novel clinic aimed at holistically serving the osteoarthritic-class III obese population for controlled and monitored weight loss through BIA.

This study is a randomized controlled trial which aims to recruit adult patients with class III obesity who present to the bariatric arthroplasty clinic. While all patients will receive individual body composition coaching to increase muscle mass and decrease body fat mass (as standard of care in this clinic), study participants will be randomly assigned to one of two cohorts: the study group who will receive nutritional and exercise consultation/intervention, or the control group who will only receive the individual body composition coaching that is standard practice at the bariatric clinic.

This study aims to identify if the addition of structured nutrition/weight loss counseling to patients at the bariatric clinic can increase the conversion from bariatric clinic to surgical candidacy from (the current) 11% to a goal of 20% by way of tracking their BIA measurements.

ELIGIBILITY:
Inclusion criteria:

* Adults, at or above 18 years of age
* BMI over 40kg/m2
* Presenting to arthroplasty-obesity clinic with desire for a total joint arthroplasty procedure

Exclusion criteria:

* Has a pacemaker or other electronic pacemaker placement
* Inability to stand unsupported for 60-90 seconds

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Weight (in kg) | 1 year
  Patient weight will be recorded at each visit
Height (in cm) | 1 year
  Patient height will be recorded at each visit
Body mass index | 1 year
  Patient BMI will be calculated by (weight in kg/height in meters squared)
Hand grip strength (measured in kg) | 1 year
  Hand grip strength will be obtained at each visit
Body fat mass | 1 year
  Body fat mass will be obtained by an InBody machine at each visit
Skeletal muscle mass | 1 year
  Skeletal Muscle mass will be obtained by an InBody machine at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States